CLINICAL TRIAL: NCT07125495
Title: The Effect of an Suction Toothbrush in Intubated Intensive Care Patients on the Development of Ventilator-Associated Pneumonia: A Randomized Controlled Trial
Brief Title: The Effect of an Suction Toothbrush on the Development of Ventilator-Associated Pneumonia
Acronym: Tootbrush_ICU
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Collaborators: Koç University Hospital (Unknown)
Responsible Party: Principal Investigator, Ayda Kebapci, Assoc Prof, Koç University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: TootbrushICU
Record Dates: First submitted 2025-08-05; First posted 2025-08-15 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Infection; Intensive Care (ICU); Intubation; Intubation Complication
Keywords: oral care; tootbrush; intensive care; intubation; Ventilatory-associated pneumonia
MeSH Terms: conditions — Infections | interventions — chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Suction tootbrush + distilled water (Experimental): All tooth surfaces, oral mucosa, and the tongue and surrounding area were cleaned every 8 hours (3x1) with distilled water and a suction toothbrush. The aspiration feature of the suction toothbrush enabled oral care and simultaneous aspiration of oropharyngeal secretions.
  Interventions: Other: Suction tootbrush and distiled water
- Suction toothbrush + 0.12% chlorhexidine gluconate oral solution (Active Comparator): Every 8 hours (3x1) 15 ml of 0.12% chlorhexidine gluconate oral solution (Adıgüzel, 2015) will be used with a suction toothbrush to clean all tooth surfaces, the oral mucosa, and the tongue. The aspiration feature of the suction toothbrush allows for the aspiration of oropharyngeal secretions during oral care.
  Interventions: Other: suction tootbrush and .12% chlorhexidine gluconate
- oral care sponge + 0.12% chlorhexidine gluconate oral solution (Active Comparator): All tooth surfaces, oral mucosa, and the tongue and surrounding tongue were cleaned with 15 ml of 0.12% chlorhexidine gluconate oral solution (Adıgüzel, 2015) every 8 hours (3x1) with an oral care sponge used in oral care.
  Interventions: Other: Oral care sponge and with 15 ml of 0.12% chlorhexidine gluconate oral solution

INTERVENTIONS:
Other: Suction tootbrush and distiled water — All tooth surfaces, oral mucosa, and the tongue and surrounding area were cleaned every 8 hours (3x1) with distilled water and a suction toothbrush. The aspiration feature of the suction toothbrush enabled oral care and simultaneous aspiration of oropharyngeal secretions.
  Arms: Suction tootbrush + distilled water
Other: suction tootbrush and .12% chlorhexidine gluconate — Every 8 hours (3x1) 15 ml of 0.12% chlorhexidine gluconate oral solution (Adıgüzel, 2015) will be used with a suction toothbrush to clean all tooth surfaces, the oral mucosa, and the tongue. The aspiration feature of the suction toothbrush allows for the aspiration of oropharyngeal secretions during oral care.
  Arms: Suction toothbrush + 0.12% chlorhexidine gluconate oral solution
Other: Oral care sponge and with 15 ml of 0.12% chlorhexidine gluconate oral solution — All tooth surfaces, oral mucosa, and the tongue and surrounding tongue were cleaned with 15 ml of 0.12% chlorhexidine gluconate oral solution (Adıgüzel, 2015) every 8 hours (3x1) and an oral care sponge used in oral care in the intensive care unit. After oral care, oropharyngeal secretions were aspirated.
  Arms: oral care sponge + 0.12% chlorhexidine gluconate oral solution

SUMMARY:
Literature suggests that suction toothbrushes may improve oral care in intubated patients by facilitating secretion removal and reducing microaspiration. This could decrease the need for endotracheal suctioning and lower the risk of ventilator-associated pneumonia (VAP). Therefore, this study aimed to examine the effect of a suction toothbrush on the development of VAP in intubated patients.

DETAILED DESCRIPTION:
in the literature examining the superiority of a suction toothbrush over another regarding the frequency of oral care practices, appropriate solution and material use in intubated patients. It is believed that a suction toothbrush will both facilitate oral care and clear oral secretions. By minimizing secretion accumulation in the mouth, it will prevent microaspiration and reduce the need for endotracheal suctioning in patients. Determining the most effective oral care method is expected to reduce the incidence of ventilator-associated pneumonia and positively impact patient mortality. Considering all this information, the aim of this study was to examine the effect of a suction toothbrush on the development of ventilator-associated pneumonia in intubated patients.

ELIGIBILITY:
Inclusion Criteria:

Patients

* who aged over 18 years
* who underwent orotracheal intubation after admission to the ICU,
* who had no known pneumonia or diagnosis of pneumonia at the time of intubation,
* who were intubated for more than 48 hours,
* who had no microorganisms detected in the tracheal aspirate within the first 48 hours,
* who had no lesions on the oral mucous membrane before intubation,
* who had no known allergy to chlorhexidine were included in the study.

Exclusion Criteria:

Patients

* who under 18 years of age,
* those with a tracheostomy,
* those were intubated for less than 48 hours,
* those with microorganisms detected in their tracheal aspirate within the first 48 hours,
* those who underwent reintubation,
* those were pregnant,
* those with lesions in the oral mucosa during intensive care admission,
* those with bleeding coagulation disorders or thrombocytopenia,
* those admitted to intensive care from an external institution while intubated, and those with a known chlorhexidine allergy were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
The ventilatory associated pneumonia (VAP) | Patients were included 48 hours after admission to the intensive care unit and intubation. After 48 hours of intubation, the development of VAP will be considered as a positive.
  The development of ventilator-associated pneumonia (VAP) after entubation in the intensive care unit (Yes / no). If a patient presents signs and symptoms of VAP with both clinical Findings and laboratory findings, researchers will diagnose it as a VAP.

CONTACTS AND LOCATIONS:
Locations (1):
- Koç University hospital Intensive care unit, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No